CLINICAL TRIAL: NCT03224429
Title: Comparative Effectiveness of a Decision Aid for Therapeutic Options in Sickle Cell Disease
Brief Title: Sickle Cell Disease (SCD) Decision Aid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Lakshmanan Krishnamurti, Proffesor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00076096
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decisional Needs Assessment (Other): Caregivers and patients with sickle cell disease will participate in a semi-structured open ended interview regarding treatment decision making.
  Interventions: Other: Qualitative Interviews Decisional Needs Assessment
- Beta Testing (Other): Caregivers and patients with sickle cell disease will review the web-based Sickle Cell Decision Aid.
  Interventions: Other: Sickle Cell Decision Aid

INTERVENTIONS:
Other: Qualitative Interviews Decisional Needs Assessment — Subjects will participate in an open-ended interview regarding type of sickle cell disease, complications, current treatment, and experiences with decision making and sickle cell treatment. Participants will be asked to describe what is important when making health care decisions. Treatment options (hydroxyurea, chronic or monthly blood transfusions, and bone marrow transplantation) will be discussed as well as how a web-based decision aid tool should be developed. The interview will be audio recorded and will take 45 to 60 minutes to complete.
  Arms: Decisional Needs Assessment
Other: Sickle Cell Decision Aid — Participants will be asked to navigate the Sickle Cell Decision Aid site that provides information about risks and benefits of therapies. As the participant navigates the site, the interviewer will ask the participants to describe thoughts about the site, including but not limited to ease of navigation, content and construction. Testing may be performed in-person or via telephone. Interviews will be audio recorded and take up to 60 to 90 minutes to complete.
  Arms: Beta Testing

SUMMARY:
The purpose of this study is to gather decision making needs information from caregivers and patients with sickle cell disease (SCD) in order to develop a web-based decision aid tool. Study subjects will participate in interviews defining treatment decision making needs during which investigators will ask information about their SCD. Notes taken from these interviews will allow the research team to better understand current practice related to clinical practice and allow for better refinement of the decision aid tool.

An additional group of participants will be asked to review the web-based Sickle Cell Decision Aid. Participants will be asked to describe thoughts about the site, including but not limited to ease of navigation, content and construction.

This study will provide information for the conduct of a randomized controlled trial for the use of a web based decision aid to give patients with sickle cell disease and parent/legal guardian of children with sickle cell disease accurate information about risks and benefits of therapies and enable them to make decisions based on their individual values and preferences.

DETAILED DESCRIPTION:
The purpose of this study is to understand patient, family and caregiver needs when making a decision about treatment for their sickle cell disease (SCD). Investigators are developing a decision aid tool that can help people understand SCD treatment options.

One group of subjects will participate in qualitative interviews defining treatment decision making needs during which investigators will ask information about their SCD. Investigators will also discuss treatment choices: hydroxyurea, chronic or monthly blood transfusions and bone marrow transplantation. Participants will be asked their thoughts about how to develop a web-based decision aid tool. Notes taken from these interviews will allow the research team to better understand current practice related to clinical practice and allow for better refinement of the decision aid tool.

An additional group of subjects will review the web-based Sickle Cell Decision Aid. Participants will be asked to navigate the site. As the participant navigates the site, the study interviewer will ask the participants to describe thoughts about the site, including but not limited to ease of navigation, content and construction. Testing may be performed in-person or via telephone. Using qualitative data collection methods, questions will be analyzed allowing for increased focus of questions based on common themes and issues identified during ongoing analysis.

This study will provide information for the conduct of a randomized controlled trial for the use of a web based decision aid to give patients with sickle cell disease and parent/legal guardian of children with sickle cell disease accurate information about risks and benefits of therapies and enable them to make decisions based on their individual values and preferences.

ELIGIBILITY:
Inclusion Criteria:

-Individual diagnosed with sickle cell disease (SCD) or parent/legal guardian/caregiver of individual (of any age) diagnosed with SCD

Exclusion Criteria:

There are no exclusions to study participation.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-03-31 (Actual)

PRIMARY OUTCOMES:
Patient/Caregiver Knowledge of Treatment Risks | Up to 90 Minutes
  Patient and caregiver knowledge of treatment risks will be collected via an open-ended semi- structured interview and aggregated as qualitative data to identify common knowledge gaps.
Patient/Caregiver Knowledge of Treatment Benefits | Up to 90 Minutes
  Patient and caregiver knowledge of treatment benefits will be collected via an open-ended semi- structured interview and aggregated as qualitative data to identify common knowledge gaps.
Patient/Caregiver Treatment Expectations | Up to 90 Minutes
  Patient and caregiver treatment expectations will be collected via an open-ended semi- structured interview and aggregated as qualitative data to identify common knowledge gaps.
Barriers to Understanding Treatment Options | Up to 90 Minutes
  Patient and caregiver knowledge of treatment options will be collected via an open-ended semi- structured interview and aggregated as qualitative data to identify common knowledge gaps.

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmanan Krishnamurti, MD, Principal Investigator — Emory University

REFERENCES:
- [Derived] Krishnamurti L, Ross D, Sinha C, Leong T, Bakshi N, Mittal N, Veludhandi D, Pham AP, Taneja A, Gupta K, Nwanze J, Matthews AM, Joshi S, Vazquez Olivieri V, Arjunan S, Okonkwo I, Lukombo I, Lane P, Bakshi N, Loewenstein G. Comparative Effectiveness of a Web-Based Patient Decision Aid for Therapeutic Options for Sickle Cell Disease: Randomized Controlled Trial. J Med Internet Res. 2019 Dec 4;21(12):e14462. doi: 10.2196/14462. PMID 31799940